CLINICAL TRIAL: NCT07090408
Title: The Effect of Chatgpt Usage on Case Analysis and Medical Artificial Intelligence Readiness Among Nursing Students: A Randomized Controlled Trial
Brief Title: Use of Artificial Intelligence in Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Yağmur AKBAL DEMİRCİ, PhD, Faculty of Health Sciences, Nursing department, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: RTEU-SBF-YAD-02
Record Dates: First submitted 2025-07-05; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Artificial Intelligence
Keywords: artificial intelligence; nursing students; nursing care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): The control arm - control group (30 students); students were asked to analyze the case with the traditional method.
- Intervention arm (Experimental): Artificial intelligence support
  Interventions: Behavioral: Artificial intelligence support

INTERVENTIONS:
Behavioral: Artificial intelligence support — Each student in the intervention group will be asked to solve a given case example using ChatGPT support. However, students in the control group will be asked to analyze the case using their own academic knowledge without ChatGPT support.
  Arms: Intervention arm

SUMMARY:
In this study, the effect of using ChatGPT, one of the artificial intelligence tools, on nursing students' case analysis and readiness for medical artificial intelligence will be evaluated.

DETAILED DESCRIPTION:
In studies on artificial intelligence in the field of nursing; it is observed that nurses reduce their workload by remotely monitoring psychiatric patients with an artificial intelligence-based sensor, there is a significant decrease in emergency room visits with an artificial intelligence-supported camera monitoring system to prevent dementia patients from falling, and the risk of pressure sores in patients in the intervention group is reduced by developing a network measurement system to predict pressure sores. Such widespread use of artificial intelligence in the nursing profession contributes to faster analysis and active management of the care process by nurses in diagnosing possible risk factors and solving any problems encountered. Thus, nurses' workload will decrease and a more efficient nursing care process will emerge. The attitude towards artificial intelligence in nursing students preparing for the profession is actually positive even in the first years of education. These results show that new generation nurses adopt artificial intelligence and its usability in the profession in the future. In fact, more academic and practical studies are needed on artificial intelligence, which has entered all professional lives in a new and rapid way. The increase in such studies, especially among students preparing for the nursing profession, will reflect both the knowledge gap in students and the necessity of proven studies in the field. The attitudes of nursing students towards new technologies and their acceptance of these innovations are especially important because they play a key role in health care. Therefore, it is necessary to learn how nursing students understand and adopt new technologies such as artificial intelligence-based technologies. When looking at the literature, it is possible to come across different studies on artificial intelligence in nursing students. However, in this study, the effect of using ChatGPT, one of the artificial intelligence tools, on case analysis and medical artificial intelligence readiness in nursing students will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Students who agree to participate in the study
* 2nd year students who are actively studying in the Nursing Department of the Faculty of Health Sciences of a university
* Students who use smartphones

Exclusion Criteria:

* Not accepting to participate in the research,
* Not using a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Case analysis delivery time | (one lesson duration) approximately 30-40 minutes
  The case analysis score was evaluated between 0 and 100 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University Faculty of Health Sciences, Rize, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I am currently undecided as I am considering this study quantitatively as well as forward-looking.